CLINICAL TRIAL: NCT00084149
Title: A Randomized Phase II Study of the Safety, Immunologic, and Virologic Effects of Cyclosporine A in Conjunction With Trizivir(R) and Kaletra(R) Versus Trizivir(R) and Kaletra(R) Alone During Primary HIV-1 Infection
Brief Title: Cyclosporine A in Combination With Abacavir Sulfate, Lamivudine, and Zidovudine and Lopinavir/Ritonavir in HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIN501/A5216; 10023 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2004-06-07; First posted 2004-06-08 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2018-08

CONDITIONS: HIV Infections
Keywords: Acute Infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; abacavir, lamivudine, and zidovudine drug combination; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporin (Experimental): Cyclosporin arm (Arm A) will receive one tablet of Abacavir sulfate, Lamivudine, and Zidovudine (ABC/3TC/AZT) twice daily, 3 capsules or 2 tablets of lopinavir/ritonavir (LPV/r) twice daily, and liquid cyclosporin A (CsA) (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Interventions: Drug: Abacavir sulfate, Lamivudine, and Zidovudine; Drug: Lopinavir/Ritonavir
- No Cyclosporin (Experimental): The No Cyclosporin arm (Arm B) will receive one tablet of Abacavir sulfate, Lamivudine, and Zidovudine (ABC/3TC/AZT) twice daily and 3 capsules or 2 tablets of lopinavir/ritonavir (LPV/r) twice daily for all 48 weeks
  Interventions: Drug: Abacavir sulfate, Lamivudine, and Zidovudine; Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine, and Zidovudine — antiretroviral therapy
  Other Names: Trizivir
Drug: Lopinavir/Ritonavir — antiretroviral therapy
  Other Names: Kaletra

SUMMARY:
Cyclosporine A (CsA) is a common long-term treatment used to inhibit the immune response in transplant patients who receive donor organs. CsA may also help people with HIV. The purpose of this study is to determine the safety of and immune response to CsA when given with abacavir sulfate (ABC), lamivudine (3TC), and zidovudine (AZT), (ABC/3TC/AZT) and lopinavir/ritonavir (LPV/r) to HIV infected adults in the early stages of infection.

Study hypothesis: The combination of CsA and LPV/r given to acutely infected individuals will result in lower levels of proviral DNA and latent infectious virus at 48 weeks compared to acute infected individuals treated with LPV/r alone.

DETAILED DESCRIPTION:
During the early stages of HIV infection, HIV replicates unchecked, massive numbers of cluster of differentiation 4 (CD4) T cells are infected and destroyed, and other CD4 cells become infected but enter a latent phase. This latent pool of infected CD4 cells poses a difficult challenge in eliminating HIV infection during the early stages of infection because the cells persist for long periods, even with highly active effective antiretroviral therapy, and may later become active.

CsA is popularly used as a lifelong immunosuppressant for organ transplant patients. CsA inhibits cellular activation, including CD4 cell activation and proliferation. By reducing CD4 cell activation during acute HIV infection, fewer CD4 cells may be infected and die; more importantly, there may be fewer latent cells with the potential to become active later in the disease. However, CsA has many potential toxic effects, including renal damage, and may affect neurologic, endocrine, and hepatic organ systems.

In a previous small study of adults with acute HIV infection, a short 8-week course of CsA was well tolerated, and it is thought that a 4-week course of CsA may result in substantial reduction in both viral load and T cell activation, outweighing any potential toxic effects sustained during the one month treatment. This study will evaluate the safety of and immune response to a 4-week course of CsA with ABC/3TC/AZT and LPV/r compared to ABC/3TC/AZT and LPV/r alone in patients with acute HIV infection.

This 48-week study will randomly assign patients to one of two arms. During the first 4 weeks of the study, Arm A will receive one tablet of ABC/3TC/AZT twice daily, 3 capsules or 2 tablets of LPV/r twice daily, and liquid CsA (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r. Arm B will receive one tablet of ABC/3TC/AZT twice daily and 3 capsules or 2 tablets of LPV/r twice daily for all 48 weeks. On a case-by-case basis, an investigator may wish to prescribe ABC/3TC rather than ABC/3TC/AZT at initial therapy. Participants with ABC hypersensitivity will be given 3TC/AZT instead of ABC/3TC/AZT.

A complete physical exam and medical history assessment will occur at study entry and at Week 48. Study visits will occur every week until Week 4, then every 4 weeks until the end of the study. Blood and urine collection and clinical assessments will occur at each study visit. Additionally, patients in Arm A only will undergo CsA level monitoring at Day 3 and Weeks 1, 2, and 3; CsA dosage may be adjusted as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Acute HIV infection with HIV viral load of more than 50,000 copies/ml AND either negative ELISA OR Western blot with 5 bands or less within 4 weeks prior to study entry
* Hepatitis B surface antigen negative within 12 weeks prior to study entry
* Hepatitis C antibody negative within 12 weeks prior to study entry
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* Prior antiretroviral therapy. A patient who has undergone Post Exposure Prophylaxis (PEP) taken at least 6 months prior to study entry is not excluded.
* Allergy or hypersensitivity to any study medications or their components
* Require certain medications, including those that may alter CsA levels or cause renal dysfunction. More information on this criterion can be found in the protocol.
* Any medical or psychiatric condition, including alcohol or drug abuse, that may interfere with adherence to study requirements
* Weight less than 88 lbs (40 kg)
* Uncontrolled hypertension
* History of pancreatitis
* History of cancer. Participants with cancer in remission who have not had treatment for at least 3 years may be eligible for this study.
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Study Chair — Aaron Diamond AIDS Research Center; Susan Little, MD, Study Chair — Department of Medicine, University of California at San Diego
Locations (4):
- United States (4):
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - MetroHealth CRS, Cleveland, Ohio

REFERENCES:
- [Background] Ravot E, Lisziewicz J, Lori F. New uses for old drugs in HIV infection: the role of hydroxyurea, cyclosporin and thalidomide. Drugs. 1999 Dec;58(6):953-63. doi: 10.2165/00003495-199958060-00001. PMID 10651384
- [Background] Rizzardi GP, Harari A, Capiluppi B, Tambussi G, Ellefsen K, Ciuffreda D, Champagne P, Bart PA, Chave JP, Lazzarin A, Pantaleo G. Treatment of primary HIV-1 infection with cyclosporin A coupled with highly active antiretroviral therapy. J Clin Invest. 2002 Mar;109(5):681-8. doi: 10.1172/JCI14522. PMID 11877476
- [Background] Rizzardi GP, Lazzarin A, Pantaleo G. Potential role of immune modulation in the effective long-term control of HIV-1 infection. J Biol Regul Homeost Agents. 2002 Jan-Mar;16(1):83-90. PMID 12003181

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclosporine: The Cyclosporine arm (Arm A) will receive one tablet of abacavir sulfate (ABC), lamivudine (3TC), and zidovudine (AZT), (ABC/3TC/AZT) twice daily, 3 capsules or 2 tablets of lopinavir/ritonavir (LPV/r) twice daily, and liquid cyclosporin A (CsA) (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
- No Cyclosporine: The No Cyclosporine arm (Arm B) will receive one tablet of ABC/3TC/AZT twice daily and 3 capsules or 2 tablets of LPV/r twice daily for all 48 weeks
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Period: Overall Study
Arm/Group | Cyclosporine | No Cyclosporine
Started | 36 | 18
Completed | 28 | 13
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- A: Cyclosporine: Arm A will receive one tablet of ABC/3TC/AZT twice daily, 3 capsules or 2 tablets of LPV/r twice daily, and liquid CsA (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
- B: Placebo: Arm B will receive one tablet of ABC/3TC/AZT twice daily and 3 capsules or 2 tablets of LPV/r twice daily for all 48 weeks
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
- Total: Total of all reporting groups
Arm/Group | A: Cyclosporine | B: Placebo | Total
Number analyzed (Participants) | 28 | 13 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [30 to 40] | 35 [30 to 43] | 36 [30 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 27 | 13 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 10 | 30
  Hispanic | 8 | 1 | 9
  African American | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 13 | 41
Cluster of differentiation 4 (CD4+) T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 407 [340 to 587] | 490 [399 to 623] | 450 [365 to 605]
Plasma log10 HIV viral load [Median (Inter-Quartile Range); unit: log10(copies/mL)] | 5.0 [4.9 to 5.8] | 4.9 [4.5 to 5.8] | 5.0 [4.7 to 5.8]

OUTCOME MEASURES:

1. Primary Outcome: Levels of Proviral DNA in Peripheral Blood Mononuclear Cells (PBMC) (log10)
Time Frame: At 48 weeks after the start of treatment
Population: All participants completing week 48 visit.
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Groups:
- Cyclosporine: Cyclosporine arm (Arm A) will receive one tablet of Abacavir sulfate, Lamivudine, and Zidovudine (ABC/3TC/AZT) twice daily, 3 capsules or 2 tablets of Lopinavir/Ritonavir (LPV/r) twice daily, and liquid Cyclosporine A (CsA) (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
- No Cyclosporine: No Cyclosporine arm (Arm B) will receive one tablet of Abacavir sulfate, Lamivudine, and Zidovudine (ABC/3TC/AZT) twice daily and 3 capsules or 2 tablets of Lopinavir/Ritonavir (LPV/r) twice daily for all 48 weeks
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
log10(copies/mL) | 1.88 [1.57 to 2.40] | 1.92 [1.77 to 2.11]

2. Secondary Outcome: Adverse Events Related to Study Medication
Description: Grade 1-4 adverse events related to study medication
Time Frame: Up to 48 weeks
Measure: Number; unit: participants
Groups:
- Cyclosporine: Cyclosporine arm (Arm A) will receive one tablet of ABC/3TC/AZT twice daily, 3 capsules or 2 tablets of LPV/r twice daily, and liquid CsA (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
- No Cyclosporine: No Cyclosporine arm (Arm B) will receive one tablet of ABC/3TC/AZT twice daily and 3 capsules or 2 tablets of LPV/r twice daily for all 48 weeks
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
participants | 1 | 0

3. Secondary Outcome: Proviral DNA Levels (log10)
Time Frame: At Week 24
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
log10(copies/mL) | 2.12 [1.71 to 2.41] | 1.96 [1.73 to 1.96]

4. Secondary Outcome: Proviral DNA (log10)
Time Frame: At Week 12
Measure: Median (Inter-Quartile Range); unit: log10(copies/mL)
Groups:
- Cyclosporine: Cyclosporine arm will receive one tablet of ABC/3TC/AZT twice daily, 3 capsules or 2 tablets of LPV/r twice daily, and liquid CsA (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
log10(copies/mL) | 2.22 [1.81 to 2.52] | 2.13 [1.97 to 2.27]

5. Secondary Outcome: HIV-1 Viral Load Levels
Time Frame: At Week 48
Measure: Mean (95% Confidence Interval); unit: log10(copies/mL)
Groups:
- No Cyclosporine: No Cyclosporine arm will receive one tablet of ABC/3TC/AZT twice daily and 3 capsules or 2 tablets of LPV/r twice daily for all 48 weeks
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
log10(copies/mL) | 1.70 [0 to 1.70] | 1.70 [0 to 1.70]

6. Secondary Outcome: Number of Patients With Viral Load Less Than 50 Copies/ml
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
Participants | 27 | 13

7. Secondary Outcome: CD4 T Cell Levels
Time Frame: At Week 48
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Cyclosporine | No Cyclosporine
Number analyzed (Participants) | 28 | 13
cells/mm^3 | 301 [146 to 432] | 287 [222 to 422]

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Groups:
- Cyclosporine: Cyclosporine will receive one tablet of ABC/3TC/AZT twice daily, 3 capsules or 2 tablets of LPV/r twice daily, and liquid CsA (dose determined by weight) twice daily. At Week 5, Arm A patients will stop CsA but continue both ABC/3TC/AZT and LPV/r.
  Abacavir sulfate, Lamivudine, and Zidovudine: antiretroviral therapy
  Lopinavir/Ritonavir: antiretroviral therapy
Arm/Group | Cyclosporine | No Cyclosporine
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/18
Other Adverse Events (participants affected / at risk) | 1/36 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclosporine (N=36) | No Cyclosporine (N=18)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No